CLINICAL TRIAL: NCT03746652
Title: A Phase 2, Multicenter, Open-label, Single-Arm Study to Evaluate the Safety and Efficacy of Daratumumab in Combination With Ixazomib and Dexamethasone as Second Line Therapy in Multiple Myeloma Patients Who Have Received Prior Treatment With a Lenalidomide Based Regimen
Brief Title: Safety and Efficacy of Daratumumab in Combination With Ixazomib and Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Acronym: DARIA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hellenic Society of Hematology (Other)
Collaborators: Janssen Pharmaceutica NV (Unknown); Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ΕΑΕ-2018/ΜΜ03
Record Dates: First submitted 2018-11-13; First posted 2018-11-20 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Multiple Myeloma
Keywords: Second line treatment; Daratumumab; Ixazomib; Dexamethasone;
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; ixazomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DId (Experimental): Daratumumab, Ixazomib, Dexamethasone
  Interventions: Drug: Daratumumab, Ixazomib, Dexamethasone

INTERVENTIONS:
Drug: Daratumumab, Ixazomib, Dexamethasone — Daratumumab 16 mg/kg, Ixazomib 4 mg, Dexamethasone 40 mg

SUMMARY:
This study will assess the efficacy of daratumumab in combination with ixazomib and dexamethasone as second line treatment for relapsed Multiple Myeloma patients.

DETAILED DESCRIPTION:
This is a Phase 2, single-arm study of daratumumab in combination with ixazomib and dexamethasone as second line treatment for relapsed Multiple Myeloma patients initially treated with lenalidomide-based regimens. Daratumumab is a human IgG1ĸ monoclonal antibody that binds with high affinity to a unique epitope on CD38, a transmembrane glycoprotein. It is a targeted immunotherapy that attacks tumor cells that overexpress CD38, in a variety of hematological malignancies including multiple myeloma. Ixazomib is an orally administered proteasome inhibitor with anti-myeloma activity.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at least 18 years of age.
2. Voluntary written informed consent before performance of any study-related procedure.
3. Relapsed patients with measurable disease parameters according to the IMWG:

   * IgG multiple myeloma: Serum M-protein level ≥1.0 g/dL or urine M-protein level ≥200 mg/24 hours, or
   * IgA, IgD, IgE, IgM multiple myeloma: Serum M-protein level ≥0.5 g/dL or urine M-protein level ≥200 mg/24 hours; or
   * Light chain multiple myeloma, for patients without measurable disease in the serum or urine: Serum immunoglobulin FLC ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda FLC ratio.
4. Patients who have received one prior regimen for MM based on lenalidomide (induction followed by any planned high dose therapy or consolidation or maintenance would be considered as one regimen).
5. Patients must have documented evidence of PD based on the investigator's determination of response as defined by the modified IMWG criteria.
6. Willingness and ability to participate in study procedures.
7. Patient has a Karnofsky Performance Status ≥ 70.
8. For patients experiencing toxicities resulting from previous therapy, the toxicities must be resolved or stabilized to ≤ Grade 1.
9. Patients with adequate bone marrow reserve, as evidenced by:

   1. Absolute neutrophil count (ANC) ≥ 1.0×10^9/L.
   2. Platelet count ≥ 75×10^9/L for patients in whom < 50% of bone marrow nucleated cells are plasma cells and ≥ 50×10^9/L for patients in whom ≥ 50% of bone marrow nucleated cells are plasma cells (transfusions are not permitted to reach this level).
10. All of the following results during Screening:

    1. Hemoglobin level ≥8 g/dL (≥ 4.65 mmol/L) (transfusions are not permitted to reach this level).
    2. Creatinine clearance ≥30 mL/min by CKD-EPI.
    3. Alanine aminotransferase (ALT) level ≤ 2.5 times the upper limit of normal (ULN).
    4. Aspartate aminotransferase (AST) level ≤ 2.5×ULN.
    5. Total bilirubin level ≤ 1.5×ULN, (except for Gilbert Syndrome: direct bilirubin ≤1.5×ULN).
    6. Serum calcium corrected for albumin ≤ 14.0 mg/dL (≤ 3.5 mmol/L), or free ionized calcium ≤ 6.5 mg/dL (≤ 1.6 mmol/L).

Exclusion Criteria:

1. Previous exposure to anti-CD38 antibodies or ixazomib.
2. Systemic treatment with or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort within 14 days before C1D1.
3. Patient has received anti-myeloma treatment within 2 weeks or 5 pharmacokinetic half-lives of the treatment, whichever is longer, prior to C1D1. The only exception is emergency use of a short course of corticosteroids (equivalent of dexamethasone 40 mg/day for a maximum of 4 days) for palliative treatment before C1D1.
4. Previous allogenic stem cell transplant; or autologous stem cell transplantation (ASCT) within 12 weeks before C1D1.
5. Patient has received radiotherapy within 14 days of C1D1. Urgent localized radiotherapy for Spinal Cord Compression is allowed.
6. History of malignancy (other than MM) within 3 years before C1D1 (exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, or other noninvasive lesion that in the opinion of the investigator, with concurrence with the Sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years).
7. Clinical signs of meningeal involvement of MM.
8. Patient has clinically significant cardiac disease, including: unstable angina or myocardial infarction within 6 months to C1D1, NYHA Class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless patient has a pacemaker, or ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) > 470 msec.
9. Known active hepatitis A, B, or C.
10. Known HIV infection.
11. Patient has a history of significant neurological, endocrine, gastrointestinal, respiratory, or inflammatory illness or stroke; or COPD requiring > 2 hospitalizations in the preceding 12 months from C1D1.
12. Patient has plasma cell leukemia (> 2.0×10^9/L circulating plasma cells by standard differential) or Waldenström's macroglobulinemia or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) or amyloidosis.
13. Patient has uncontrolled hypertension or hypertension requiring >2 medications for adequate control within 14 days to C1D1.
14. Patient has uncontrolled diabetes within 14 days to C1D1 or diabetes mellitus with > 2 episodes of ketoacidosis in the preceding 12 months from C1D1.
15. Patient has ongoing ≥ Grade 2 peripheral neuropathy.
16. Patient had ≥ Grade 3 rash during prior therapy.
17. Patient has had major surgery within 14 days prior to C1D1, or has not fully recovered from an earlier surgery, or has surgery planned during the time the patient is expected to participate in the study or within 2 weeks after the last dose of study drug administration. Note: patients with planned surgical procedures to be conducted under local anesthesia may participate. Kyphoplasty or vertebroplasty are not considered major surgery.
18. Pregnant or nursing women.
19. Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence.
20. Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.
21. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
22. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
23. Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | From first day of treatment until end of study, documented progressive disease (PD), or death (approximately up to 36 months)
  ORR is defined as the proportion of patients who achieve a best response of PR or better, using modified IMWG criteria.

SECONDARY OUTCOMES:
Evaluation of the hematologic and non-hematologic toxicity profile of the combination. | From first day of treatment until end of study, PD, or death (approximately up to 36 months)
  Toxicities related to the administration of Daratumumab or Ixazomib will be assessed (e.g., neutropenia, thrombocytopenia, nausea, peripheral neuropathy, rash, etc.).
Duration of response (DOR) | From the date of initial documentation of a response (CR, VGPR or PR) to the date of first documented evidence of PD, as defined in the IMWG criteria (approximately up to 36 months)
  For patients who have not progressed, data will be censored at the last disease evaluation before the start of any subsequent anti-myeloma therapy.
Time to disease progression (TTP) | From C1D1 to the date of first documented evidence of PD, as defined in the IMWG criteria (approximately up to 36 months)
  Time in months from first dose of treatment until PD.
Progression-free survival (PFS) | From C1D1 to either PD, according to the IMWG criteria, or death, whichever occurs first (approximately up to 36 months)
  For patients who have not progressed and are alive, data will be censored at the last disease evaluation before the start of any subsequent anti-myeloma therapy. Relapse from CR by positive immunofixation or trace amount of M-protein is not considered to be PD and is not included in the PFS calculation.
Overall survival (OS) | From C1D1 to the date of death from any cause (approximately up to 36 months)
  Overall survival (OS) is measured from C1D1 to the date of the patient's death. If the patient is alive or the vital status is unknown at the time of the analysis, then the patient's data will be censored at the date the patient was last known to be alive.
Time to next therapy (TNT) | From C1D1 to the date of the next anti-neoplastic therapy or death from any cause, whichever comes first (approximately up to 36 months)
  For patients who neither start a new anti-neoplastic therapy nor die, survival time will be censored at the date of their last available follow-up date. For a patient who does not have any post-baseline follow-up assessments and who has not died, survival time will be censored at C1D1.
Minimal Residual Disease (MRD) negativity using Next-Generation Flow Cytometry (NGFC) | Assessed every 3 months post CR/sCR until PD (approximately up to 36 months)
  MRD negativity rate is defined as the proportion of patients who achieve a negative result of MRD. Patients without MRD assessment will be considered as having MRD-positive results.
Serum bone markers | The evaluation will be performed on C1D1 and then every 3 months until PD (approximately up to 36 months)
  NTX, CTX, bALP, RANKL, OPG, Dkk-1, SOST and serum angiogenic cytokines levels angiogenin, VEGF, angiopoietin-1 and -2.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Terpos, Prof., Principal Investigator — Department of Clinical therapeutics, National and Kapodistrian University of Athens, School of medicine, Athens, Greece
Locations (1):
- General Hospital of Athens "Alexandra", Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No